CLINICAL TRIAL: NCT02388321
Title: Comparison of Sub-dissociative Dose Intranasal Ketamine to Intranasal Fentanyl for Treatment of Moderate to Severe Pain in Pediatric Patients Presenting to the Emergency Department: a Prospective, Randomized, Double-blind Study
Brief Title: Pediatric Ketamine Study for Pain Management
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients meeting inclusion criteria was low, and PI went to another institution.
Sponsor: Antonios Likourezos (Other)
Collaborators: Maimonides Medical Center (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-11-20-MMC
Record Dates: First submitted 2015-02-09; First posted 2015-03-17 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: Analgesia; pediatrics; pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): intranasal sub-dissociative dose ketamine for the treatment of moderate to severe pain in pediatric patients in the emergency department.
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): intranasal fentanyl for the treatment of moderate to severe pain in pediatric patients in the emergency department.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — intranasal sub-dissociative dose ketamine for the treatment of moderate to severe pain in pediatric patients in the emergency department.
  Arms: Ketamine
Drug: Fentanyl — intranasal fentanyl for the treatment of moderate to severe pain in pediatric patients in the emergency department.
  Other Names: Fetanyl
  Arms: Fentanyl

SUMMARY:
Direct comparison of intranasal sub-dissociative dose ketamine with intranasal fentanyl for the treatment of moderate to severe pain in pediatric patients in the emergency department.

DETAILED DESCRIPTION:
Intranasal (IN) delivery of analgesic agents provides rapid and convenient drug administration without the need for needles. In children, the placement of an intravenous line often increases anxiety and pain, requires nursing time, and can be very difficult to achieve, so the IN route is particularly advantageous. IN delivery of fentanyl has become increasingly more common in pain management for children in many settings, including pre-hospital and emergency department (ED) settings. Over the past decade, many studies have demonstrated that intranasal fentanyl is as effective as intravenous morphine to treat acute moderate to severe pain. Intranasal fentanyl has become standard of care in some pediatric EDs with the advantage of avoiding intravenous line placement. However, adverse effects attributed to IN fentanyl are similar to those of other opioid analgesics: hypotension, sedation, and occasionally respiratory depression. Ketamine is a noncompetitive N-methyl D-aspartate (NMDA) receptor antagonist that blocks the release of the excitatory neurotransmitter glutamate and provides anesthesia, amnesia, and analgesia by decreasing central sensitization and "wind-up" phenomenon. Due to its high lipid solubility, ketamine rapidly crosses the blood-brain barrier, provides rapid onset of action (peak concentration at 1 minute after intravenous push) and rapid recovery to baseline (duration of action 5-15 minutes after intravenous push). At sub-dissociative doses, either used as an adjunct to opioid analgesics or as a solo agent, ketamine provides effective analgesia while preserving airway patency, ventilation, and cardiovascular stability.

Ketamine has been less studied for pain management, however it has been safely used via different routes of administration in children. Studies dating back to 1990's use ketamine at doses as high as 6 mg/kg intranasally in children for pre-medication prior to surgery or for sedation with little or no reported adverse effects. A hospital in Australia is currently conducting a clinical trial comparing IN fentanyl 1.5 ug/kg to IN ketamine 1mg/kg for the treatment of pain caused by isolated musculoskeletal injury. The intention of our study is similar to this, however the investigators will not limit the patients to those with only musculoskeletal pain and a more simplified pain scale will be used.

To assess pain, the investigators will use the standard pain scale that is currently used in our Pediatric ED in order to minimize the need to re-train any of our staff with a different pain scale. The scale incorporates the Numerical rating scale (0-10 scale; NRS) and the Wong-Baker faces pain scale (6 faces corresponding to 0,2,4,6,8,10; WBS). While prior studies have used different pain scales, primarily the visual analog scale (VAS), the scales that the investigator currently use have been validated in children in 2009.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-17,
* weighing less than 50kg
* present to the pediatric ED with moderate-severe acute pain (defined as pain greater than or equal to 6/10).
* Treating physician determines the patient to require opioid analgesia.

Exclusion Criteria:

* Children with facial trauma or any abnormal nasal anatomy;
* developmentally delayed children;
* children with head trauma/increased intracranial pressure (ICP);
* children with known allergy to fentanyl or ketamine;
* children who are unable to provide pain scale assessment;
* children with chronic pain of greater than 4 weeks;
* Pregnant females;
* and children with a Glasgow Coma Scale (GCS)<15.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Zavolkovskaya, MD, Principal Investigator — Maimonides Medical Center; Sergey Motov, MD, Study Director — Maimonides Medical Center; John Marshall, MD, Study Chair — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Background] Borland ML, Clark LJ, Esson A. Comparative review of the clinical use of intranasal fentanyl versus morphine in a paediatric emergency department. Emerg Med Australas. 2008 Dec;20(6):515-20. doi: 10.1111/j.1742-6723.2008.01138.x. PMID 19125831
- [Background] Borland M, Milsom S, Esson A. Equivalency of two concentrations of fentanyl administered by the intranasal route for acute analgesia in children in a paediatric emergency department: a randomized controlled trial. Emerg Med Australas. 2011 Apr;23(2):202-8. doi: 10.1111/j.1742-6723.2011.01391.x. Epub 2011 Feb 8. PMID 21489168
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Goldman RD: Intranasal drug delivery for children with acute illness. Curr Drug Ther 2006, 1(1):127-130.
- [Background] Grassin-Delyle S, Buenestado A, Naline E, Faisy C, Blouquit-Laye S, Couderc LJ, Le Guen M, Fischler M, Devillier P. Intranasal drug delivery: an efficient and non-invasive route for systemic administration: focus on opioids. Pharmacol Ther. 2012 Jun;134(3):366-79. doi: 10.1016/j.pharmthera.2012.03.003. Epub 2012 Mar 23. PMID 22465159
- [Background] Graudins A, Meek R, Egerton-Warburton D, Seith R, Furness T, Chapman R. The PICHFORK (Pain InCHildren Fentanyl OR Ketamine) trial comparing the efficacy of intranasal ketamine and fentanyl in the relief of moderate to severe pain in children with limb injuries: study protocol for a randomized controlled trial. Trials. 2013 Jul 10;14:208. doi: 10.1186/1745-6215-14-208. PMID 23842536
- [Background] Holdgate A, Cao A, Lo KM. The implementation of intranasal fentanyl for children in a mixed adult and pediatric emergency department reduces time to analgesic administration. Acad Emerg Med. 2010 Feb;17(2):214-7. doi: 10.1111/j.1553-2712.2009.00636.x. PMID 20070272
- [Background] Karlsen AP, Pedersen DM, Trautner S, Dahl JB, Hansen MS. Safety of intranasal fentanyl in the out-of-hospital setting: a prospective observational study. Ann Emerg Med. 2014 Jun;63(6):699-703. doi: 10.1016/j.annemergmed.2013.10.025. Epub 2013 Nov 22. PMID 24268523
- [Background] Miner JR, Kletti C, Herold M, Hubbard D, Biros MH. Randomized clinical trial of nebulized fentanyl citrate versus i.v. fentanyl citrate in children presenting to the emergency department with acute pain. Acad Emerg Med. 2007 Oct;14(10):895-8. doi: 10.1197/j.aem.2007.06.036. PMID 17898251
- [Background] National Institute of Clinical Studies: Emergency care acute pain management manual, National Health and Medical Research Council. Canberra, Australia: ACT; 2011.
- [Background] Page MG, Katz J, Stinson J, Isaac L, Martin-Pichora AL, Campbell F. Validation of the numerical rating scale for pain intensity and unpleasantness in pediatric acute postoperative pain: sensitivity to change over time. J Pain. 2012 Apr;13(4):359-69. doi: 10.1016/j.jpain.2011.12.010. Epub 2012 Mar 15. PMID 22424915
- [Background] Rickard C, O'Meara P, McGrail M, Garner D, McLean A, Le Lievre P. A randomized controlled trial of intranasal fentanyl vs intravenous morphine for analgesia in the prehospital setting. Am J Emerg Med. 2007 Oct;25(8):911-7. doi: 10.1016/j.ajem.2007.02.027. PMID 17920976
- [Background] Saunders M, Adelgais K, Nelson D. Use of intranasal fentanyl for the relief of pediatric orthopedic trauma pain. Acad Emerg Med. 2010 Nov;17(11):1155-61. doi: 10.1111/j.1553-2712.2010.00905.x. PMID 21175512
- [Background] Yeaman F, Meek R, Egerton-Warburton D, Rosengarten P, Graudins A. Sub-dissociative-dose intranasal ketamine for moderate to severe pain in adult emergency department patients. Emerg Med Australas. 2014 Jun;26(3):237-42. doi: 10.1111/1742-6723.12173. Epub 2014 Apr 8. PMID 24712757
- [Background] Yeaman F, Oakley E, Meek R, Graudins A. Sub-dissociative dose intranasal ketamine for limb injury pain in children in the emergency department: a pilot study. Emerg Med Australas. 2013 Apr;25(2):161-7. doi: 10.1111/1742-6723.12059. Epub 2013 Mar 20. PMID 23560967

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Fentanyl
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Fentanyl | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.5) | 9.6 (2.9) | 9.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 30 Minutes
Description: An 11 point Likert Visual Analog Scale with 0 being no pain, 5 being moderate pain and 10 being very severe pain was verbally administered to the patient at 30 minutes post administration of analgesia.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 11 | 11
units on a scale | 3.36 (2.6) | 2.09 (2.3)

2. Secondary Outcome: Adverse Events at 30 Minutes
Description: The patient were asked at 30 minutes post administration of analgesia if they experienced any side effects like nausea, vomiting, headache etc.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketamine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=11) | Fentanyl (N=11)
Dizzines (Nervous system disorders) | 5 (5) | 1 (1) — Dizziness

LIMITATIONS AND CAVEATS:
Small Sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No